CLINICAL TRIAL: NCT02330744
Title: The Neurobiology of Approach Avoidance Training in Depression
Acronym: ACTIV8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Charles Taylor, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21695
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Approach-positive AAT (Experimental): Computerized AAT procedure designed to increase automatic approach responses for positive social cues.
  Interventions: Behavioral: Approach-positive AAT
- Control AAT (Placebo Comparator): Computerized AAT procedure in which there is no contingency between arm movement and positive social cues.
  Interventions: Behavioral: Control AAT

INTERVENTIONS:
Behavioral: Approach-positive AAT — One session of approach-positive AAT (Aim 1 and 2) followed by 4 sessions of approach-positive AAT over 2 weeks concurrent with a brief computer-delivered behavioral activation treatment for depression (Aim 3).
  Arms: Approach-positive AAT
Behavioral: Control AAT — One session of control-AAT (Aim 1 and 2) followed by 4 sessions of control-AAT over 2 weeks concurrent with a brief computer-delivered behavioral activation treatment for depression (Aim 3).
  Arms: Control AAT

SUMMARY:
The purpose of this study is to test the effects of a computerized approach/avoidance training (AAT) procedure on behavioral, affective, and brain mechanisms that are important for reward sensitivity and well-being in individuals diagnosed with major depression. The training procedure is designed to modify automatic approach responses for positive social stimuli. The primary aim is to determine the effects of approach/avoidance training on the functioning of brain systems during reward processing in individuals diagnosed with major depression. A secondary aim will determine whether brain activation patterns following approach/avoidance training predict subsequent affective and behavioral responses during reward processing. An exploratory aim will test whether completing the approach/avoidance training procedure in combination with a brief computer-delivered behavioral activation program for depression will produce larger changes in depression symptoms, positive emotions, and social relationship functioning from pre- to post-intervention compared to the control training procedure.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55
* Principal psychiatric diagnosis of major depressive disorder
* Patient Health Questionnaire - 9 item score ≥ 10
* Ability to read and speak English sufficiently to complete study procedures

Exclusion Criteria:

* History of psychosis, mania, or substance dependence
* Current severe medical disorder that requires inpatient treatment or frequent medical follow ups including but not limited to: unstable hypertension, unstable angina, unstable diabetes mellitus, unstable cardiac arrhythmias, transient ischemic attacks, sever coronary artery disease, sever peripheral vascular disease, severe hepato-gastro-intestinal disease, severe infectious disease (e.g. HIV), recurrent severe headache or migraine, fainting spells, seizures, and history of traumatic brain injury with loss of consciousness > 30 minutes
* Current use of the following medications: antidepressants, benxodiazepines, antipsychotics, mood stabilizers, or other drugs that can acutely affect the hemodynamic response (methylphenidate and acetazolamide)
* Caffeine intake > 10 cups/day or recent significant changes in consumption
* MRI exclusions, including claustrophobia, cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a metal worker/welder, history of eye surgery/eyes washed out because of metal, women who are or may be pregnant (determined by a positive pregnancy test), women using an intrauterine device, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; older tattoos with metal dyes; unwillingness to remove nose, ear, tongue or face rings.
* Concurrent psychosocial treatment: Participants completing ongoing psychosocial treatment will be required to meet a 12-week stability criteria so that symptom changes as a result of other psychosocial treatments are not confounded with changes due to the research.
* Inability to complete the initial assessment battery or behavioral training sessions.
* Clinical conditions assessed by the interviewer that necessitate more imminent clinical care (e.g., active suicidal ideation). These criteria are in place so participants with these other, more several symptoms can be referred for appropriate mental health services.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change from pre-training in blood oxygen level dependent (BOLD) response in the striatum, amygdala, and medial prefrontal cortex, as measured with functional magnetic resonance imaging (fMRI) during reward trials on the Social Incentive Delay (SID) task. | Post-training (5 minutes)
  Change from pre- to post-training in neural activation during social reward processing.

SECONDARY OUTCOMES:
Response bias to rewards on the Probabilistic Reward Task (PRT) | Post-training (20 minutes) and 1 month
  Post-training (20 minutes; Aim 2) and post-AAT plus brief behavioral activation treatment (1 month; Aim 3) reward response bias on the PRT.
Response to social interaction task | Post-training (30 minutes) and 1 month
  Post-training (30 minutes; Aim 2) and post-AAT plus brief behavioral activation treatment (1 month; Aim 3) behavioral and emotional response to the social interaction task.

OTHER OUTCOMES:
Change from baseline in depression (Patient Health Questionnaire-9; Beck Depression Inventory II, composite) | 1 month
  Change from pre- to post-assessment following AAT plus brief behavioral activation treatment (Aim 3) in symptoms of depression.
Change from baseline in positive affect (Positive and Negative Affect Schedule) | 1 month
  Change from pre- to post-assessment following AAT plus brief behavioral activation treatment (Aim 3) in positive affect.
Change from baseline in social relationship functioning (Social Connectedness Scale - Revised; Interpersonal Outcomes Scale) | 1 month
  Change from pre- to post-assessment following AAT plus brief behavioral activation treatment (Aim 3) in social relationship functioning.
Change from baseline in anhedonia (Mood and Symptom Anxiety Questionnaire; Environmental Reward Observation Scale) | 1 month
  Change from pre- to post-assessment following AAT plus brief behavioral activation treatment (Aim 3) in anhedonia.
Change from baseline in anxiety (State Trait Anxiety Inventory). | 1 month
  Change from pre- to post-assessment following AAT plus brief behavioral activation treatment (Aim 3) in anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Charles T Taylor, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego; Psychiatry Clinical Research, San Diego, California, United States

REFERENCES:
- [Derived] Bomyea J, Choi SH, Sweet A, Stein M, Paulus M, Taylor C. Neural Changes in Reward Processing Following Approach Avoidance Training for Depression. Soc Cogn Affect Neurosci. 2021 Oct 13;17(3):336-49. doi: 10.1093/scan/nsab107. Online ahead of print. PMID 34643736